CLINICAL TRIAL: NCT06359860
Title: A Phase Ib/II Study to Evaluate the Efficacy and Safety of ST-1898 in Subjects With Unresectable or Metastatic Melanoma
Brief Title: A Study of ST-1898 for Unresectable or Metastatic Melanoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Scitech-Mq Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ST-1898-203
Record Dates: First submitted 2024-01-03; First posted 2024-04-11 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Unresectable or Metastatic Melanoma
Keywords: ST-1898; Melanoma
MeSH Terms: conditions — Melanoma | interventions — 3-(3'-adamantan-1-yl-4'-methoxybiphenyl-4-yl)-2-propenoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ST-1898 Phase Ib (Experimental): Dose Escalation: Subjects will be administered orally at 140mg, 160mg, 180mg, 220mg, QD during the study, until disease progression or intolerable toxicity.
  Interventions: Drug: ST-1898 tablets
- ST-1898 Phase II (Experimental): Dose Expansion: Subjects with unresectable or metastatic melanoma will be administered orally at recommended phase II dose from phase Ib once daily during the study, until disease progression or intolerable toxicity.
  Interventions: Drug: ST-1898 tablets

INTERVENTIONS:
Drug: ST-1898 tablets — Supplied as 5 mg and 40 mg tablets

SUMMARY:
ST-1898 is a receptor tyrosine kinase (RTK) inhibitor for multi-targets, especially for VEGFR2, c-MET, AXL, PDGFRA, RET, KIT etc. This trial is to evaluate its safety, tolerability, pharmacokinetic, and efficacy in subjects with unresectable or metastatic melanoma.

In phase Ib, the primary objectives are to assess the safety and tolerability, and to determine Recommended Phase 2 dose (RP2D) of ST-1898 tablets in subjects with unresectable or metastatic melanoma. Secondary objectives are to assess the plasma concentration of ST-1898 and to evaluate the efficacy.

In phase II, the primary objective is to assess the anti-tumor activities of ST-1898 tablets in subjects with unresectable or metastatic melanoma. The secondary objective is to evaluate the safety of ST-1898 tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Life expectancy of three months or more
3. Histologically or cytologically confirmed unresectable or metastatic stage III or IV acral melanoma that was progressed with conventional therapy
4. Recommendation of subject offering archived tissue sample or previous biomarker test report. If archived tumor sample is not available, a fresh biopsy is optional, which need to be taken from needle biopsy or core needle biopsy (fine needle biopsy not allowed)
5. Eastern Cooperative Oncology Group performance status (PS) ≤ 1
6. At least one measurable lesion per RECIST 1.1
7. Has adequate organ function defined as follows:

   * Absolute neutrophil count ≥ 1.5 ×10^9/L, Platelets ≥ 75× 10^9/L and Hemoglobin ≥ 90 g/L (no blood transfusions, no platelet transfusions and no use of colony stimulating factor within 2 weeks prior to routine blood test) at screening;
   * Serum creatinine ≤1.5 × upper limit of normal (ULN)
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 ULN, AST/ALT ≤ 5 ULN for liver metastasis;
   * Total bilirubin ≤ 1.5 ULN
   * International normalized ratio (INR) ≤ 1.5 ULN, or prothrombin time (PT) ≤1.5 ULN
   * Activated partial thromboplastin time (APTT) ≤1.5 ULN
   * Serum albumin ≥30 g/L
8. Willing and able to provide written Informed consent.
9. Eligible male and female subjects with fertility activity or their sexual partners must use effective contraception during study period and though 90 days after last study treatment. Women of child-bearing age must have a negative serum pregnancy test within 7 days before first study treatment

Exclusion Criteria

1. Subjects with one of the following conditions prior to first dose, including, but not limiting to：

   * A history of antitumor therapy within 4 weeks, including chemotherapy, radiotherapy, biotherapy, endocrine therapy or immunotherapy, etc.;
   * A history of oral fluoropyrimidines and small molecular targeted-drug therapy within 2 weeks or 5 half-life time （the longer time taken as final）;
   * A history of traditional Chinese medicine with antitumor indication within 2 weeks;
2. A history of being participant in clinical trial of other unapproved drugs within 4 weeks;
3. A major operation or severe trauma within 4 weeks, （except tumor biopsy, puncture,）invasive dental procedures such as dental extraction, dental implants etc.
4. Current or previous severe retinopathy who, in the judgment of the Investigator, are not suitable for enrollment
5. A history of clinically significant cardiovascular or cerebrovascular disease, including, but not limiting to:

   * Severe arrhythmia or heart conduction disturbance, such as second-degree or third-degree atrio-ventricular block or ventricular arrhythmia indicated with medical intervention
   * QTc (by Fridericia): male >450 ms, female >470 ms
   * Major cardiovascular events within 6 months prior to first dose, including acute coronary syndrome, stroke, deep vein thrombosis, pulmonary-thromboembolism and other ≥Grade 3 arterial-thrombosis events, or congestive heart failure, or aortic dissection etc.；
   * New York Heart Association Class ≥ II；
   * Left ventricular ejection fraction（LVEF）<50%；
   * Uncontrolled hypertension (blood pressure≥140/90 mmHg even with antihypertensive therapy)
6. Subjects with active leptomeningeal disease or brain metastases without being well controlled, except subjects with asymptomatic or treated brain metastases being stable imaging between 12 weeks before screening；
7. Subjects with interstitial lung disease or radiation pneumonia in needs of corticosteroids therapy
8. Subjects with clinically uncontrolled pleural effusion, pericardial effusion, or ascites requiring frequent drainage or medical intervention within 7 days prior to first dose;
9. Subjects with malignant tumors in the last 5 years (not including non-melanoma skin cancer, breast cancer or cervical cancer in situ, and superficial bladder transient cell carcinoma that have been cured)
10. A history of ≥ grade 3 bleeding episodes within 6 months prior to first dose; or currently ≥ grade 2 hemorrhage, with angioneoplasm/ vascular malformation, with high bleeding risks (such as active peptic ulcer or esophageal varices)
11. Within 2 weeks prior to first dose of concomitant medication with strong inducers of CYP3A4, strong inhibitors of CYP3A4, or substrates with narrow therapeutic windows of CYP3A4;
12. Subjects with ≥ Grade 2 (by CTCAE) toxicities caused by previous therapy (not including ≤Grade 2 peripheral neuropathy, alopecia, or other tolerated and no possible safety hazard events as determined by the investigator);
13. Subjects with active hepatitis B, unless HBV-DNA titer in the normal range (for subjects with positive HBsAg but HBV-DNA titer eligible, prophylactic antiviral therapy except interferon is allowed); active hepatitis C (ANTI-HCV positive)；
14. Subjects with positive HIV antibodies or Treponema pallidum antibodies;
15. Subjects with acute bacterial, viral or fungal infections, and in needs of systemic antimicrobial therapy;
16. Pregnant or lactating females;
17. Subjects with significant neuropsychiatric disorders, leading to poor compliance;
18. Subjects with underlying diseases (including abnormal laboratory investigations), alcohol, drug abuse, or drug dependence, all which affect the interpretation of toxicities or adverse event, or decrease;
19. Subjects with oral administration impossible, or in the conditions of malabsorption as determined by the investigator, such as dysphagia and intestinal obstruction, etc.;
20. Subjects with significant liver cirrhosis, hepatatrophy, portal hypertension, or more than moderate volume of ascites;
21. A history of organ transplant;
22. A history of other severe systemic disease, or not suitable as determined by the investigator due to any other reasons;
23. A history of inoculation with live vaccine within 28 days prior to first dose. Note: Seasonal influenza vaccine is a broadly inactivated vaccine and is permitted. Inactivated COVID-19 vaccines are permitted. COVID-19 mRNA vaccines are not allowed. Intranasal influenza vaccines are live vaccines and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ib Dose Escalation: The Number and frequency of treatment-related adverse events (AEs) and treatment related serious adverse events (SAEs) | Approximately 18 months
  AEs and SAEs will be assessed according to the National Cancer Institute (NCI) CTCAE v5.0
Phase Ib Dose Escalation: Recommended Phase 2 Dose (RP2D) | Within the first cycle (21days)
  RP2D was determined according to MTD. MTD was defined as the highest dose level at which no more than 1 in 6 participants experienced a dose-limiting toxicity (DLT) during the first cycle (21days) of treatment.
Phase II Expansion: Objective Response Rate (ORR) | Approximately 18 months
  ORR is defined as the percentage of participants who experience a CR or PR based on RECIST 1.1 (CR: Complete Response, Disappearance of all target lesions, PR: Partial Response, At least a 30% decrease in the sum of diameters of target lesions)

SECONDARY OUTCOMES:
Phase Ib Dose Escalation: Trough concentration of ST-1898 | Cycle 1 Day 1, Cycle 1 Day 21, Cycle 3 Day 1 during Phase Ib Dose Escalation (21 days per cycle), up to 10 weeks
  To assess plasma pharmacokinetics (PK) of oral administration of ST-1898
Phase Ib Dose Escalation: Peak concentration of ST-1898 | Cycle 1 Day 1, Cycle 1 Day 21, Cycle 3 Day 1 during Phase Ib Dose Escalation (21 days per cycle), up to 10 weeks
  To assess plasma pharmacokinetics (PK) of oral administration of ST-1898
Phase Ib Dose Escalation: ORR | Approximately 18 months
  Objective Response Rate (ORR) per RECIST 1.1
Phase Ib Dose Escalation: PFS | Approximately 18 months
  Progression-Free Survival (PFS) per RECIST 1.1
Phase Ib Dose Escalation: DoR | Approximately 18 months
  DoR Duration of Response (DoR) per RECIST 1.1
Phase Ib Dose Escalation: DCR | Approximately 18 months
  Disease Control Rate (DCR) per RECIST 1.1
Phase Ib Dose Escalation: TTP | Approximately 18 months
  Time to Progression per RECIST 1.1
Phase II Dose Expansion: The Number and frequency of treatment-related adverse events and serious adverse events (SAEs) | Approximately 18 months
  The AEs and SAEs will be assessed according to the National Cancer Institute (NCI) CTCAE v5.0.
Phase II Dose Expansion: Trough concentration of ST-1898 | Cycle 1 Day 1, Cycle 1 Day 21, Cycle 3 Day 1 during Phase II Dose Expansion (21 days per cycle), up to 10 weeks
  To assess plasma Trough concentration of oral administration of ST-1898 in subjects with unresectable or metastatic melanoma
Phase II Dose Expansion: Peak concentration of ST-1898 | Cycle 1 Day 1, Cycle 1 Day 21, Cycle 3 Day 1 during Phase II Dose Expansion (21 days per cycle), up to 10 weeks
  To assess plasma Peak concentration of oral administration of ST-1898 in subjects with unresectable or metastatic melanoma
Phase II Dose Expansion: PFS | Approximately 18 months
  Progression-Free Survival (PFS) per RECIST 1.1
Phase II Dose Expansion: DoR | Approximately 18 months
  DoR Duration of Response (DoR) per RECIST 1.1
Phase II Dose Expansion: DCR | Approximately 18 months
  Disease Control Rate (DCR) per RECIST 1.1
Phase II Dose Expansion: TTP | Approximately 18 months
  Time to Progression per RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jun GUO, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, China

IPD SHARING:
Plan to Share IPD: No